CLINICAL TRIAL: NCT05174520
Title: Comparative Effects of Muscle Energy Technique and Routine Physical Therapy on Quadratus Lumborum in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Comparative Effects of Muscle Energy Technique and Routine Physical Therapy on Quadratus Lumborum in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Hadia Ehsan, Principal investigator, University of Lahore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MSPTM02193012
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Chronic Low-back Pain
Keywords: Low back pain; Lumbar pain; Backache; Muscle Energy Technique; Quadratus Lumborum
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Physical Therapy group (Active Comparator): Routine physical therapy group includes thermotherapy for 10 mins, transcutaneous electrical nerve stimulations for 10 mins. Exercises such as: Pelvic tilts, bridging exercise, William flexion exercises and stretching will be performed for 7-10 repetitions.
  Treatment duration will be 25 minutes.
  Interventions: Other: Routine Physical Therapy
- Experimental group (Experimental): Experimental group includes 6-7 repetitions of Muscle energy technique on Quadratus Lumborum muscle and Routine physical therapy, i.e Thermotherapy, transcutaneous electrical nerve stimulations, Pelvic tilts, bridging exercise, William flexion exercises and stretching will be performed for 7-10 repetitions.
  Treatment duration will be 40 minutes.
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: Routine Physical Therapy — Routine physical therapy will be provided to group A for 25 minutes thrice a week for 4 weeks.
  Other Names: Conventional Physical Therapy
  Arms: Routine Physical Therapy group
Other: Muscle Energy Technique — Muscle Energy technique along with Routine physical therapy will be provided to group B for40 minutes thrice a week for 4 weeks.
  Arms: Experimental group

SUMMARY:
•Null hypothesis: There is no difference in effects of Muscle Energy Technique and Routine Physical Therapy on Quadratus Lumborum in patients with chronic low back pain.

•Alternative hypothesis: There is difference in effects of Muscle Energy Technique and Routine Physical Therapy on Quadratus Lumborum in patients with chronic low back pain.

DETAILED DESCRIPTION:
The purpose of the study is to compare the effects of Muscle Energy Technique and Routine Physical Therapy on Quadratus Lumborum in patients with chronic low back pain on Pain, Range of Motion, Quality of Life and Functional Disability.

The study procedure will be explained to the patients and informed written consent will be obtained from those patients who will be willing to participate in the study. Quadratus Lumborum tightness will be assessed using side bending test.

Those fulfilling the requirement of inclusion criteria will be indiscriminately separated into 2 groups. NPRS, Oswestry Disability Index, SF-20 and goniometer will be used to collect data.

Total 68 participants will be recruited in the study. Routine Physical therapy will be provided to group A. Reciprocal inhibition Muscle Energy Technique on quadratus lumborum along with Routine Physical Therapy will be performed on group B.

Both group will receive interventions three sessions in a week for 4 consecutive weeks.

Assessment of Pain, Range of motion, Quality of Life and Functional Disability will be assessed by using goniometer, NPRS, Oswestry Disability Index and SF-20 Questionnaire respectively for both groups at the baseline, end of 6th session (2nd week) and end of 12th session (4th week) and follow up will be obtained after 1 month (8th week).

ELIGIBILITY:
Inclusion Criteria:

* Both genders of age 30 to 55 year.
* Patients with pain for at least three months or more (chronic stage).
* Patients having score of at least 3 on 0-10 points(NPRS).
* Diagnosed patients of low back pain.
* Non-radicular low back pain.
* Quadratus Lumborum tightness by physical test i.e. side bending test.

Exclusion Criteria:

* Pregnant females.
* Lumbar radiculopathy.
* Any spinal pathology i.e. infectious disease and fracture.
* Any congenital deformity of spine, upper and lower extremities.
* Systemic illnesses i.e. cardiovascular disorders, respiratory disorders etc.
* History of surgery of hip, pelvis, lumbar spine, disc herniation.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Pain will be assessed by Numeric pain rating scale | 1 minute
  Pain will be measured using 11 point Numeric Pain rating scale (NPRS). 0 score represents no pain, 1-3 score represents mild pain, 4-6 represents moderate pain and 7-10 represents severe pain.
Range of Motion will be assessed by Universal Goniometer | 2 minutes
  Lumbar flexion, extension and side bending range of motion will be measured using Universal Goniometer. Normal lumbar flexion range is 60 degrees, extension range is 25 degrees, and right and left side bending range is 25 degrees.
Quality of life will be assessed by Medical outcomes study: 20 item Short form survey instrument | 8 minutes
  The SF-20 measure contains three dimensions about function (physical, social and role) and well-being (mental health, health perception and pain). score between 75- 100 leveled as good quality of life of low back pain patients, Average QOL marked when QOL score between 50-74, and QOL score between 0-49 leveled as poor QOL.
Functional Disability will be assessed by Oswestry Low Back Pain Disability Index | 5 minutes
  Oswestry disability index is a validated, 10-point patient-reported outcome questionnaire. • 0% to 20% is scored as minimal disability. • 21%-40% is scored as moderate disability. • 41%-60% is scored as severe disability. • 61%-80% is scored as crippled. • 81%-100% scored as bedbound patients.

CONTACTS AND LOCATIONS:
Overall Officials: M Waqar Afzal, Mphil-MSK, Study Chair — University of Lahore; Syed Asadullah Arslan, Ph.D. PT, Study Director — University of Lahore
Locations (1):
- University of Lahore teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No